CLINICAL TRIAL: NCT04461314
Title: MedPAC Hotline: A Medical Peer Addiction Counselling Hotline Service for Drug-abusing Youth and Young Adults
Brief Title: Hotline Service for Drug-abusing Youth and Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MedPAC Hotline
Record Dates: First submitted 2020-06-15; First posted 2020-07-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-07

CONDITIONS: Drug Abuse
Keywords: Youth; Hotline; Drug abuse; Young Adult; Addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-led counselling (Other): 1. About 50 university students trained as peer telephone counsellors through a structured training programme.
  2. About 200 Drug-abusing youth and young adults received telephone-based, Peer-led Brief Motivational Interviewing (BMI)
  Interventions: Behavioral: peer-led counselling

INTERVENTIONS:
Behavioral: peer-led counselling — About 50 university students will be trained as peer counsellors through a structured training programme. A pre and post and 6-month self-administered questionnaire will be conducted before, immediately and 6-month after the training programme to examine their changes of knowledge and attitudes. A satisfaction survey will also be conducted to measure participants' perception of the quality of the training programme.
  Drug-abusing youth and young adults will receive telephone-based, Peer-led Brief Motivational Interviewing (BMI) counselling to rehabilitate from drug abuse. The peer counsellors will give referral advice if the youth and young adult needs appropriate treatment and rehabilitation services.
  The drug abusers will be counselled and invited to complete the follow-up questionnaires at 1 week, 1 month, 3 months, 6 months, 9 months and 1 year. Self-reported quitters at 6-month and 1-year follow-ups will be invited to have a urine test to validate the drug abuse abstinence.

SUMMARY:
Aim: Providing peer counselling service delivered by student counsellors with a medical background via a hotline to drug-abusing youth and young adult aged 35 or below.

Objectives:

i. To raise anti-drug awareness of young people in general and identify high-risk/hidden drug-abusing youth and young adult aged 35 or below in Hong Kong; and ii. To train university students with a medical background as peer counsellors; and iii. To provide drug abuse hotline service by students with a medical background as peer counsellors to drug-abusing youth and young adult aged 35 or below, and other people who call for help, including drug abusers' family members, friends, and professionals; and iv. To improve the drug-abusing youth and young adult' knowledge about the hazard of drug abuse, negative attitude, and perception towards the drug abuse through the telephone peer counselling service provided by students with medical background; and v. To increase the intention to quit and the help-seeking behavior among the drug-abusing youth and young adult; vi. To increase reduction rate and abstinence rate from drug abuse, and decrease the relapse rate among drug-abusing youth and young adult through the telephone peer counseling service.

DETAILED DESCRIPTION:
The MedPAC Hotline Service will be promoted to high-risk and drug-abusing youth and young adults through a variety of platforms, namely schools and youth service organizations, industries, community, mass media and internet, social media, posters and snowball approach.

The hotline service will operate from 5 p.m. to 9 p.m. on weekday and from 2 p.m. to 8 p.m. on weekend. A peer counsellor or a research assistant will answer the telephone inquiries from 9:30 a.m. to 5 p.m. on weekdays.

About 50 university students will be trained as peer counsellors through a structured training programme. The students will be invited to complete the pre, post and 6-month self-administered questionnaire before, immediately and 6-month after the training programme to examine their changes of knowledge of and attitudes towards addiction counselling. A satisfaction survey will also be conducted to measure their perception on the quality of training programme.

Peer counsellors will use telephone-based, Peer-led Brief Motivational Interviewing (BMI) counselling to motivate and encourage drug-abusing or high-risk youth and young adults to rehabilitate from drug abuse, assist them to manage the withdrawal symptoms, and help identify barriers and facilitators to rehabilitate from drug abuse in the telephone counselling. The peer counsellors will give referral advices if the youth and young adult needs appropriated treatment and rehabilitation services.

The drug-abusing youth and young adults will be counselled and invited to complete the follow-up questionnaires over the telephone after joining the MedPAC Hotline Service programme for 1 week, 1 month, 3 months, 6 months, 9 months and 1 year. Self-reported quitters at 6-month and 1-year follow-ups were invited to have urine test to validate the drug abuse abstinence status.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of target service group for this quitline programme is that current drug abusers in Hong Kong who should (1) be aged 35 or below, (2) be able to communicate in Cantonese, and (3) have a history of drug abuse within the past 12 months (including all types of drugs such as narcotics analgesics, hallucinogens, depressants, stimulants, tranquillizers and other recreational drugs).
* The inclusion criteria of peer counsellors providing counselling service in this quitline programme are those who should (1) be aged 18 - 35, (2) be able to communicate in Cantonese, (3) have a medical background, (4) complete the training courses and pass the evaluation of peer counsellor qualification.

Exclusion Criteria:

* Those who are psychologically or physically unable to communicate will be excluded.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in drug consumption at 12-month follow-up | Baseline and 12 months
  Drug abuser's drug consumption is measured at 12-month follow-up. A questionnaire asking the frequency of drug use in the past 30 days will be used for assessing the self-reported change in drug consumption.

SECONDARY OUTCOMES:
30 days self-reported drug abstinence at 6-month and 12-month follow-up | Baseline, 6 months and 12 months
  Self-reported drug abstinence (do not use drug for at least 30 days during the time of follow-up) at 6-month and 12-month. A questionnaire asking the drug use status, quitting experience will be used for assessing the self-reported drug abstinence.
Change in drug consumption at 6-month follow-up | Baseline and 6 months
  Drug abuser's drug consumption is measured at 6-month follow-up. A questionnaire asking the frequency of drug use in the past 30 days will br used for assessing the self-reported change in drug consumption.
Change in relapse risk among the quitters | Baseline and 12 months
  Drug quitter's relapse risk is measured at 12-month follow-up. A questionnaire using Stimulant Relapse Risk Scale (SRRS) with the questions of the intention to use drugs, compulsivity for drugs and impetus and confidence to avoid drugs etc. will be used for assessing the relapse risk at 12-month follow-up. The higher the scores, the higher the relapse risk.
Change of the contemplation stage | Baseline, 6 months and 12 months
  Drug abuser's change of the contemplation stage at 6-month and 12-month follow-up. A questionnaire asking the intention to quit drug abuse and experience of drug abstinence to match the stage in contemplation ladder will be used for assessing the contemplation stage at 6-month and 12-month.
Changes of the perceived treatment needs and motivation towards solving the problem of drug abuse | Baseline, 6 months and 12 months
  Drug abuser's change of perceived treatment needs and motivation towards solving the problem among drug abusers at 6-month and 12-month. A questionnaire using the Treatment Needs/Motivation Scales (TCU MOTForm) will be used for assessing the level of the intention and motivation to receive treatment of solving the drug abuse problem. The higher the scores, the higher the perceived treatment needs and motivation.
Change of self-efficacy of drug abusers to avoid drug use | Baseline, 6 months and 12 months
  Drug abuser's change of self-efficacy to avoid drug use at 6-month and 12-month follow-up. The Adolescent Relapse Coping Questionnaire (ARCQ) will be used for evaluating the self-efficacy to avoid drug use. It comprises 6 questions for a given condition about drug temptation. The higher the score, the higher the self-efficacy of drug abusers to avoid drug use.
Drug abuser's improvement of knowledge and attitude on drug abuse hazards | Baseline, 6 months and 12 months
  Drug abuser's improvement of knowledge and attitude on drug abuse hazards at 6-month and 12-month follow-up. A questionnaire asking about the knowledge and attitude on drug abuse with a scale called "knowledge and attitude on drug abuse for drug abuser" will be used for assessing the change of knowledge and attitude on drug abuse. The higher the scores, the better the knowledge and attitude.
Peer counsellor's improvement of knowledge and attitude on drug abuse hazards | Baseline, immediately after the training programme and 6 months
  Peer counsellor's improvement of knowledge and attitude on drug abuse hazards immediately after the training programme and after 6 months will be measured by a scale called "knowledge and attitude on drug abuse for peer counsellor" in a self-reporting structured questionnaire. The higher the scores, the better the knowledge and attitude.
Satisfaction of peer counsellors to the drug abuse training programme | Immediately after the training programme
  Satisfaction of peer counsellors to the drug abuse training programme will be collected. A questionnaire asking about the comments of content, practicability, speakers from the peer counsellors with the satisfaction scale will be used for evaluating the satisfaction immediately after the training programme. The higher the scores, the greater the satisfaction of the training programme.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Pokfulam, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient-level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project have been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)

REFERENCES:
- [Derived] Xia W, Li HCW, Liang T, Luo Y, Ho LLK, Cheung AT, Song P. Structured online training for university students to deliver peer-led addiction counselling for young drug abusers in China: Effect on improving knowledge, attitude, confidence, and skills. Patient Educ Couns. 2022 Apr;105(4):1009-1017. doi: 10.1016/j.pec.2021.07.038. Epub 2021 Jul 24. PMID 34334262